CLINICAL TRIAL: NCT07015892
Title: Phase III Randomized Clinical Trial to Evaluate the Efficacy and Safety of Twice-Daily Hyperfractionated Dose-Escalated Thoracic Radiotherapy in Patients With Limited-Stage Small Cell Lung Cancer (ESCALADOR Study)
Brief Title: Dose-Escalation Radiotherapy in Limited-Stage Small Cell Lung Cancer: A Phase III Randomized Trial
Acronym: ESCALADOR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCALADOR Study; PI 2024 11 1761 (Registry Identifier: Ethics Committee for Clinical Research of the Health Area of Salamanca (CEIm Salamanca))
Record Dates: First submitted 2025-05-28; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Radiotherapy; Chemoradiotherapy; Dose-Response Relationship; Radiation
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Eligible patients are randomized in a 1:1:1 ratio to one of three parallel treatment arms. All arms include concurrent chemoradiotherapy with cisplatin and etoposide, but differ in the radiotherapy dose and technique: standard-dose BID radiotherapy (45 Gy), dose-escalated BID radiotherapy (60 Gy), or BID radiotherapy with a simultaneous integrated boost to 54 Gy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Radiotherapy Arm (45 Gy BID) (Active Comparator): Patients in this group will receive concurrent chemoradiotherapy consisting of cisplatin and etoposide with standard-dose thoracic radiotherapy: 45 Gy administered in 30 fractions of 1.5 Gy twice daily (BID).
  Interventions: Radiation: Thoracic Radiotherapy 45 Gy BID
- Escalated Dose Radiotherapy Arm (60 Gy BID) (Experimental): Patients in this group will receive the same chemotherapy as Arm 1, combined with an escalated thoracic radiotherapy dose: 60 Gy delivered in 40 fractions of 1.5 Gy twice daily (BID). Dose may be reduced to 54 Gy if organs at risk exceed tolerance.
  Interventions: Radiation: Thoracic Radiotherapy 60 Gy BID
- Simultaneous Integrated Boost Radiotherapy Arm (45-54 Gy BID) (Experimental): Patients in this group will receive the same chemotherapy as in other arms, with thoracic radiotherapy delivered as a simultaneous integrated boost (SIB): 45 Gy to the general target volume and 54 Gy to the high-risk clinical target volume (CTV) in 30 fractions BID.
  Interventions: Radiation: Thoracic Radiotherapy SIB 45-54 Gy BID

INTERVENTIONS:
Radiation: Thoracic Radiotherapy 45 Gy BID — 45 Gy delivered in 30 fractions of 1.5 Gy twice daily over three weeks, with 95% of the planning target volume (PTV) receiving at least 95% of the prescribed dose.
  Arms: Standard Radiotherapy Arm (45 Gy BID)
Radiation: Thoracic Radiotherapy 60 Gy BID — 60 Gy delivered in 40 fractions of 1.5 Gy BID. A minimum dose of 54 Gy will be accepted if organ-at-risk tolerance is exceeded.
  Arms: Escalated Dose Radiotherapy Arm (60 Gy BID)
Radiation: Thoracic Radiotherapy SIB 45-54 Gy BID — 45 Gy in 30 fractions (1.5 Gy BID) to PTV and 54 Gy in 30 fractions (1.8 Gy BID) to high-risk CTV. Both delivered simultaneously using 3D conformal planning.
  Arms: Simultaneous Integrated Boost Radiotherapy Arm (45-54 Gy BID)

SUMMARY:
This is a phase III clinical trial that aims to evaluate whether increasing the dose of radiotherapy given twice a day can improve treatment outcomes in patients with localized small cell lung cancer (SCLC). All patients will receive standard chemotherapy with cisplatin and etoposide and will be randomly assigned to one of three radiotherapy regimens.

The main objective is to determine whether this intensified radiotherapy improves progression-free survival and overall survival. The study will also compare two different dose escalation strategies and assess treatment side effects and patients' quality of life.

This research may help identify a more effective treatment approach for patients with limited-stage SCLC and could contribute to improving long-term survival in this aggressive type of cancer

DETAILED DESCRIPTION:
This is a phase III, prospective, randomized, multicenter trial designed to evaluate whether a dose escalation strategy using twice-daily hyperfractionated thoracic radiotherapy can improve outcomes in patients with limited-stage small cell lung cancer (LS-SCLC).

Patients will be randomly assigned to one of three treatment arms: (A) standard-dose radiotherapy (45 Gy in 30 fractions BID), (B) escalated-dose radiotherapy (60 Gy in 40 fractions BID), or (C) standard-dose with a simultaneous integrated boost (45-54 Gy BID). All patients will receive concurrent chemotherapy with cisplatin and etoposide.

The study aims to determine if intensified radiotherapy increases progression-free survival (PFS) and overall survival (OS). Secondary objectives include comparing toxicity profiles, quality of life (using EORTC QLQ-C30 and LC13/LC29), and exploratory analyses of circulating biomarkers.

LS-SCLC has high recurrence rates despite aggressive treatment. Although BID thoracic radiotherapy (TRT) of 45 Gy is considered standard, new evidence suggests that higher doses may further improve survival without increasing toxicity. Modern radiotherapy techniques and improved imaging (e.g., PET-CT) allow more accurate targeting and potential dose escalation.

The study plans to enroll 300 patients over 36 months across 10-15 Spanish centers, coordinated by the Instituto de Investigación Biomédica de Salamanca (IBSAL) and supported by SEOR-GOECP. An interim analysis will be conducted at year 1 and year 3, with a final analysis at 5 years. Data will be collected via REDCap and follow FAIR principles. The protocol has been approved by the Salamanca Research Ethics Committee.

This trial seeks to define whether a higher radiotherapy dose improves long-term outcomes in LS-SCLC and to explore how biomarker data might inform future personalized treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of small cell lung cancer (SCLC)
* Limited-stage disease (Stage I-III; any T, any N, M0), eligible for definitive radiotherapy
* Measurable disease according to RECIST 1.1
* Age ≥18 years
* ECOG performance status 0-2
* No prior thoracic radiotherapy
* Signed informed consent
* Adequate hematologic function: WBC ≥3.0×10⁹/L, neutrophils ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥90 g/L
* Adequate liver and renal function: total bilirubin ≤1.5×ULN, AST/ALT ≤1.5×ULN, creatinine normal or CrCl ≥60 mL/min
* Pulmonary function: FEV1 >1 L or >30% predicted; DLCO >30% predicted

Exclusion Criteria:

* Prior surgery or radiotherapy for any lung cancer (SCLC or NSCLC)
* Presence of malignant cells in pleural or pericardial effusion
* Serious uncontrolled systemic disorders (e.g., active infection, unstable cardiovascular disease)
* Medical, psychological, or social conditions that could interfere with compliance
* Active malignancy other than SCLC (except localized prostate/breast cancer or basal cell carcinoma)
* Refusal or inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until disease progression or death, whichever occurs first, assessed up to 5 years
  Progression-Free Survival (PFS) is defined as the time from randomization to documented disease progression based on RECIST 1.1 criteria or death from any cause. Patients will be evaluated at baseline, every 3 months for the first 2 years, then every 6 months up to year 5 using imaging and clinical assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until death from any cause, assessed up to 5 years
  Overall Survival (OS) is defined as the time from randomization to death from any cause. Patients will be followed longitudinally through scheduled clinical visits and survival status checks
Incidence of Acute and Late Toxicities (per CTCAE v4.0) | From treatment initiation through 5-year follow-up
  Toxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Both acute and late toxicities (e.g., esophagitis, pneumonitis, hematologic toxicity) will be recorded during treatment and follow-up.
Quality of Life Assessment (EORTC QLQ-C30) | Baseline, 3 months, 6 months, 12 months, and annually up to 5 years
  Quality of life will be measured using the EORTC QLQ-C30. Changes in scores over time will be analyzed to evaluate treatment impact on physical, emotional, and functional well-being. The EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) is a validated instrument designed to assess the quality of life of cancer patients. It includes 30 items organized into multi-item scales and single-item measures, covering a range of functional domains, symptoms, and overall health status. All items are scored on a 1 to 4 Likert scale (1 = "Not at all" to 4 = "Very much"), except for the two items of the global health status/QoL scale, which are scored from 1 to 7 (1 = "Very poor" to 7 = "Excellent").
  A high score on a functional scale reflects better functioning. A high score on a symptom scale reflects worse symptom severity. A high global health/QoL score indicates overall good health and quality of life as perceived by the patient.
Quality of life Assesment (LC13) | Baseline, 3 months, 6 months, 12 months, and annually up to 5 years
  Quality of life will be measured using lung cancer-specific module LC13. Changes in scores over time will be analyzed to evaluate treatment impact on physical, emotional, and functional well-being. The EORTC QLQ-LC13 is a lung cancer-specific module designed to be used in conjunction with the EORTC QLQ-C30. It focuses on lung cancer-related symptoms and treatment side effects, particularly from chemotherapy and radiotherapy. Just like with the QLQ-C30, raw scores are linearly transformed to a 0-100 scale for each item or symptom scale. Higher scores always reflect worse symptoms or more severe treatment-related side effects. A change of ≥10 points is typically considered clinically meaningful.
  Combined with the QLQ-C30, the LC13 enhances sensitivity to lung-specific disease burden and treatment toxicity.
Quality of Life Assesment (LC29) | Baseline, 3 months, 6 months, 12 months, and annually up to 5 years
  Quality of life will be measured using the lung cancer-specific module LC29. Changes in scores over time will be analyzed to evaluate treatment impact on physical, emotional, and functional well-being. The EORTC QLQ-LC29 is a lung cancer-specific quality of life questionnaire, that captures a broader and more contemporary range of lung cancer symptoms and treatment-related side effects, especially relevant to newer therapies like immunotherapy and targeted agents. The QLQ-LC29 is designed to be used in conjunction with the EORTC QLQ-C30. All items are scored on a 1-4 Likert scale:
  1. = Not at all
  2. = A little
  3. = Quite a bit
  4. = Very much Scores are linearly transformed to a 0-100 scale. For all LC29 items and scales: Higher scores indicate more severe symptoms or problems.
  LC29 retains some items from LC13 (e.g., cough, dyspnea, pain) but adds new domains (e.g., fear of progression, trouble concentrating). Provides a broader range of symptoms, including psychosocial concerns.
Time to First Local or Distant Recurrence | From randomization until first documented recurrence, assessed up to 5 years
  Time to recurrence will be measured based on clinical and radiological evaluations. Recurrences will be categorized as local (within the irradiated field) or distant (outside the thoracic field).

CONTACTS AND LOCATIONS:
Overall Officials: Iñigo San Miguel Arregui, MD PhD, Principal Investigator — Institute of Biomedical Research of Salamanca
Locations (13):
- Spain (13):
  - Complejo Asistencial Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario de Torrecardenas, Almería
  - Hospital Universitario de Cruces, Barakaldo
  - Instituto Catalán de Oncología, Girona
  - Hospital Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Marques de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Genesis Care, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in future publications (after de-identification) will be made available upon reasonable request. This includes data related to baseline characteristics, treatment administration, toxicity, tumor response, survival outcomes, and quality of life assessments
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available starting 12 months after publication of primary results and for a minimum of 5 years thereafter.
Access Criteria: Qualified researchers with a methodologically sound proposal, as determined by the study steering committee, will be able to access the data. Requests should be directed to the study PI. A data access agreement will be required